CLINICAL TRIAL: NCT06340984
Title: Role of Intercellular Adhesion Molecule -1 in Acne Vulgaris Patients : Effect of Montelukast Therapy
Brief Title: Serum Intercellular Adhesion Molecule -1 in Acne Vulgaris Patients : Effect of Montelukast
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Alshayma Gamal Fouad, doctor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sICAM-1 in acne vulgaris
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — montelukast; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group moderate acne (Active Comparator): patients with moderate acne vulgaris who will receive Montelukast therapy dose: 10mg/day, duration of therapy: three months, serum level of intercellular adhesion molecule -1 will be measured by performing an enzyme-linked immune sorbent assay (E LISA) before and after treatment
  Interventions: Drug: Montelukast 10 Mg Oral Tablet
- group severe acne (Active Comparator): patients with severe acne vulgaris who will receive Montelukast therapy dose: 10mg/day, duration of therapy: three months, serum level of intercellular adhesion molecule -1 will be measured by performing an enzyme-linked immune sorbent assay (E LISA) before and after treatment
  Interventions: Drug: Montelukast 10 Mg Oral Tablet
- control group (No Intervention): Healthy patients with Age and sex matching ,No history of acne, serum level of intercellular adhesion molecule -1 will be measured by performing an enzyme-linked immune sorbent assay (E LISA)

INTERVENTIONS:
Drug: Montelukast 10 Mg Oral Tablet — group modrate and severe acne will receive Montelukast therapy , dose: 10mg/day, duration of therapy: three months., Quantitively assay of level of serum intercellular adhesion molecule -1 will be measured by performing an enzyme-linked immune sorbent assay (E LISA) in group moderate acne vs group severe acne pre Montelukast treatment and after three months of treatment vs control group
  Other Names: level of serum intercellular adhesion molecule -1 will be measured by performing an enzyme-linked immune sorbent assay (E LISA)
  Arms: group moderate acne; group severe acne

SUMMARY:
The aim of this study is to:

1. Evaluation of serum soluble intercellular adhesion molecule-1 (sICAM-1) level in acne vulgaris and compare it to control group
2. Evaluate its role in acne pathogenesis and its correlation with acne vulgaris severity
3. Evaluate the effect of Montelukast on serum (sICAM-1) level in acne vulgaris

DETAILED DESCRIPTION:
Acne vulgaris is a common chronic skin disease involving blockage and inflammation of pilosebaceous units

. It is characterized by non-inflammatory, open or closed comedones and by inflammatory lesions include papules, pustules and nodules. Affecting mostly the face, but also the back and chest .

Acne vulgaris may have a psychological impact on any patient, regardless of the severity or the grade of the disease .

Prevalence of self-reported acne was 34.7%. Females significantly reported acne more frequently than males (39.1% vs. 30.3%) Prevalence of clinically confirmed acne was 24.4%, with higher rates among females (28.6%) than males (20.2%).

Its pathogenesis result from increased sebum production (due to increased activity of androgens and insulin growth factor-1), excessive deposition of keratin in pilosebaceous follicles leading to comedo formation, colonization of the follicle by Propionibacterium acnes bacteria, and the local release of pro-inflammatory chemicals in the skin through certain inflammatory mechanisms.

Recently, Inflammation is a key feature in the pathogenesis of acne vulgaris, with various chemokines and cytokines that contribute to fuel a vicious cycle .

Leukotriene B4 (LT-B4) is the most potent leucocyte chemotactic mediator in the pathogenesis of acne . Intercellular adhesion molecule-1 (ICAM-1) is a transmembrane glycoprotein in the immunoglobulin superfamily that increases in response to various inflammation mediator, In addition, genetics is also a key factor in the pathophysiology of acne .

There are various topical therapies for acne vulgaris including topical retinoids, antimicrobials, benzoyl peroxide, salicylic acid, lactic acid, dapsone and niacinamide. Moderate to severe acne is treated with oral antibiotics, especially tetracyclines, and isotretinoin is prescribed for severe acne unresponsive to antibiotics.

Montelukast is an antagonist of LT-B4 receptor . Montelukast has good efficacy, tolerability, and safety in the treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons of both sexes with moderate and severe acne vulgaris.
* Patients age between 15-35 years
* Patients with acne vulgaris not receiving any topical or systemic treatments for acne at least 2 weeks and 2 month before the study ,respectively

Exclusion Criteria:

* Pregnant and lactating women
* Diabetics
* Hypertensive patients
* acne conglobate patients and acne fulminans patients
* patients with history of polycystic ovaries syndrome
* Patients with history of thyroid dysfunction
* Patients with history of chronic inflammatory or immune-mediated diseases as Crohn's disease, vascular dementia, systemic sclerosis, systemic lupus erythematosus, ankylosing spondylitis, psoriatic arthritis and SAPHO syndrome.
* Any history of hypersensitivity reaction to the studied drug

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of serum soluble intercellular adhesion molecule-1 (sICAM-1) level in acne vulgaris (moderate -severe ) | baseline and three months at the end of treatment
  evaluation of serum soluble intercellular adhesion molecule-1 (sICAM-1) level by ELISA in acne vulgaris(moderate -severe) and compare it to control group, correlation with acne vulgaris severity and its role in pathogenesis
Montelukast in treatment of acne vulgaris patients | three months following end of treatment
  Evaluate the effect of Montelukast on serum (sICAM-1) level in acne vulgaris (group moderate acne vs group severe acne )and its side effects

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Mohammed Ibrahim, Assistant Professor, Study Director — South Valley University; Abdulrahman Abdul Hamid Alsaied, Professor, Study Director — South Valley University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hazarika N. Acne vulgaris: new evidence in pathogenesis and future modalities of treatment. J Dermatolog Treat. 2021 May;32(3):277-285. doi: 10.1080/09546634.2019.1654075. Epub 2019 Aug 29. PMID 31393195
- [Background] Kellett SC, Gawkrodger DJ. The psychological and emotional impact of acne and the effect of treatment with isotretinoin. Br J Dermatol. 1999 Feb;140(2):273-82. doi: 10.1046/j.1365-2133.1999.02662.x. PMID 10233222
- [Background] Tayel K, Attia M, Agamia N, Fadl N. Acne vulgaris: prevalence, severity, and impact on quality of life and self-esteem among Egyptian adolescents. J Egypt Public Health Assoc. 2020 Nov 5;95(1):30. doi: 10.1186/s42506-020-00056-9. PMID 33165744
- [Background] Goulden V, McGeown CH, Cunliffe WJ. The familial risk of adult acne: a comparison between first-degree relatives of affected and unaffected individuals. Br J Dermatol. 1999 Aug;141(2):297-300. doi: 10.1046/j.1365-2133.1999.02979.x. PMID 10468803
- [Background] Borgia F, Peterle L, Custurone P, Vaccaro M, Pioggia G, Gangemi S. MicroRNA Cross-Involvement in Acne Vulgaris and Hidradenitis Suppurativa: A Literature Review. Int J Mol Sci. 2022 Mar 17;23(6):3241. doi: 10.3390/ijms23063241. PMID 35328662
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Background] Roebuck KA, Finnegan A. Regulation of intercellular adhesion molecule-1 (CD54) gene expression. J Leukoc Biol. 1999 Dec;66(6):876-88. doi: 10.1002/jlb.66.6.876. PMID 10614768
- [Background] Rokni GR, Mohammadnezhad F, Saeedi M, Shadi S, Sharma A, Sandhu S, Gupta A, Goldust M. Efficacy, tolerability, and safety of montelukast versus finasteride for the treatment of moderate acne in women: A prospective, randomized, single-blinded, active-controlled trial. J Cosmet Dermatol. 2021 Nov;20(11):3580-3585. doi: 10.1111/jocd.14462. Epub 2021 Oct 14. PMID 34648685
- [Background] Grice CA, Tays KL, Savall BM, Wei J, Butler CR, Axe FU, Bembenek SD, Fourie AM, Dunford PJ, Lundeen K, Coles F, Xue X, Riley JP, Williams KN, Karlsson L, Edwards JP. Identification of a potent, selective, and orally active leukotriene a4 hydrolase inhibitor with anti-inflammatory activity. J Med Chem. 2008 Jul 24;51(14):4150-69. doi: 10.1021/jm701575k. Epub 2008 Jun 28. PMID 18588282
- [Background] Zouboulis CC, Bettoli V. Management of severe acne. Br J Dermatol. 2015 Jul;172 Suppl 1:27-36. doi: 10.1111/bjd.13639. PMID 25597508
- [Background] Del Rosso JQ. Oral Doxycycline in the Management of Acne Vulgaris: Current Perspectives on Clinical Use and Recent Findings with a New Double-scored Small Tablet Formulation. J Clin Aesthet Dermatol. 2015 May;8(5):19-26. PMID 26029331
- [Background] Alestas T, Ganceviciene R, Fimmel S, Muller-Decker K, Zouboulis CC. Enzymes involved in the biosynthesis of leukotriene B4 and prostaglandin E2 are active in sebaceous glands. J Mol Med (Berl). 2006 Jan;84(1):75-87. doi: 10.1007/s00109-005-0715-8. Epub 2005 Dec 31. PMID 16388388
- See also: 2. Mustafa S A G. An Overview About Acne Vulgaris. Journal of Pharmaceutical Negative Results.(2022):4395-4402 — https://scholar.google.com/scholar?hl=ar&as_sdt=0%2C5&q=2.%09Mustafa+S+A+G.+An+Overview+About+Acne+Vulgaris.+Journal+of+Pharmaceutical+Negative+Results.%282022%29%3A4395-4402+&btnG=
- See also: 14. U.S. Department of Health and Human Services Food and Drug Administration Center for Drug Evaluation and Research (CDER).Guidance for industry. Acne vulgaris: developing drugs for treatment.(2005). — http://www.fda.gov/regulatory-information/search-fda-guidance-documents/acne-vulgaris-establishing-effectiveness-drugs-intended-treatment